CLINICAL TRIAL: NCT01228253
Title: Effects of Treatment of Post-traumatic Stress Disorder on Reduced Recall for Fear Extinction
Brief Title: Effects of Treatment of PTSD on Reduced Recall for Fear Extinction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-PP-05
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (No Intervention): Safe voluntary.
- 2 (No Intervention): patient with psychotrauma but without PSTD and without any psychiatric trouble at the time of inclusion
- 3 (No Intervention): patient with psychotrauma and PTSD (post-traumatic stress disorder) and in full remission at the time of inclusion
- 4.3 (No Intervention): patient with psychotrauma and with activ PTSD (post-traumatic stress disorder)at the time of inclusion
- 4.2 (Sham Comparator): patient with psychotrauma and with activ PTSD (post-traumatic stress disorder)at the time of inclusion
  Interventions: Device: SHAM rTMS: repetitive transcranial magnetic stimulation is off
- 4.1 (Experimental): patient with psychotrauma and with activ PTSD (post-traumatic stress disorder)at the time of inclusion
  Interventions: Device: rTMS: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: rTMS: repetitive transcranial magnetic stimulation — patients will be treated with rTMS at 10 Hz (D3 to D7 and D10-D14, 1 session / day)
  Arms: 4.1
Device: SHAM rTMS: repetitive transcranial magnetic stimulation is off — patients will be treated with rTMS at 10 Hz (D3 to D7 and D10-D14, 1 session / day with the stimulator on off
  Other Names: SHAM rTMS: repetitive transcranial magnetic stimulation
  Arms: 4.2

SUMMARY:
This preliminary study will examine the differential effects of rTMS on the recall of extinction of conditioned fear in patients suffering from PTSD (post-traumatic stress disorder ) compared with subjects without PTSD but with high risk of relapse.

DETAILED DESCRIPTION:
It is estimated that nearly 70% of individuals will experiment at least once in their life a traumatic event (eg war, natural disaster, accident or assault). The psychotrauma, whose symptoms (including revivalism, hypersensitivity to the environment, anxiety, avoidance behavior), may be sustainable and thus constitute a posttraumatic stress disorder (PTSD). One characteristic of PTSD can be studied in the laboratory is the lack of recall of extinction of conditioned fear, caused largely by a lack of induction of hyperactivation in the prefrontal cortex. Knowing that this hyperactivation may occur in some cases of remission of symptoms of PTSD, it is possible that the deficit in recall of extinction is lifted in such cases. This idea is also supported by animal models showing that the induction of natural or artificial prefrontal hyperactivation facilitates the recall of extinction. However, no study has yet addressed so far the effects of different treatments (conventional: pharmacotherapy and psychotherapy, or rTMS: repetitive transcranial magnetic stimulation) for PTSD, supposed to induce prefrontal hyperactivation and avoid the recall deficit of extinction of conditioned fear. The persistence of this deficit beyond the remission of PTSD symptoms could represent a situation with a high risk of relapse.

Objective. Our main objective is to examine performance in recall of extinction of conditioned fear on the one hand, in patients in remission of PTSD after conventional treatment and, secondly, in patients who received rTMS at 10 Hz

Population: THIS PRELIMINARY STUDY will include 9 patients with PTSD, 3 individuals in remission from PTSD, 3 psychotraumatized subjects without secondary PTSD and 3 individuals without a history of psychotrauma. These groups will be matched for age, sex and sociocultural level.

Method: All studies will be conducted at the Nice University Hospital. The pre-inclusion visit (D-7), including different clinical evaluations (MINI-DSM-IV, CAPS, PDI, Hamilton Depression Scale and Covi Anxiety), will be held at the Emergency Psychiatric Unit (Hospital Saint-Roch). The study will take place at the Psychiatry University Department and at the Neurology Exploration Department (Hospital Pasteur), where the subjects will have other clinical assessments (at D0, D17-D19, D21), the conditioning test and extinction (day 0) and recall test of extinction (at D21). The fear conditioning (measured by increases in heart rate and skin conductance) corresponds to presentations coupled with an image and tactile stimulation (the intensity of which will be chosen by the subject), while sessions of extinction and extinction recall that correspond to presentations of the image alone (without tactile stimulation). In addition to these sessions, one third of PTSD patients will be treated with rTMS at 10 Hz (D3 to D7 and D10-D14, 1 session / day), another third with placebo treatment and one third without treatment. Eventually (D21), two other tests will indirectly assess prefrontal hyperactivation (emotional Stroop and attentional bias) and self-questionnaires will be performed in all subjects immediately after the recall of extinction.

The persistent failure to recall extinction in some individuals in remission from PTSD would sign the maintenance of prefrontal dysfunction, and therefore a high risk of relapse. The induction of hyperactivation using prefrontal rTMS at 10 Hz would not only reduce symptoms of PTSD, but also reduce the risk of recurrence of these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* French mother tongue
* major
* patient out of hospital
* patient with health insurance

Exclusion Criteria:

* patient with dysthymia
* alcohol dependence, drug dependence
* acute or chronic psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
prefrontal hyperactivation | Day 21
  recall test of extinction (at D21)

SECONDARY OUTCOMES:
neuropsychological tests | Day 21
  two other tests will indirectly assess prefrontal hyperactivation (emotional Stroop and attentional bias)

CONTACTS AND LOCATIONS:
Overall Officials: Michel BENOIT, PhD, Principal Investigator — psychiatry department, Nice University Hospital
Locations (1):
- Chu de Nice, Nice, France